CLINICAL TRIAL: NCT00064727
Title: Attenuating Insulin Resistance as a Therapeutic Target in the Management of Heart Failure
Brief Title: Rosiglitazone to Treat Patients With Heart Failure and Glucose Intolerance or Type II Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030217; 03-H-0217
Record Dates: First submitted 2003-07-10; First posted 2003-07-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-04-11

CONDITIONS: Congestive Heart Failure
Keywords: Ventricular Contractile Function; Diastolic Dysfunction; PPAR gamma; Gene Expression Patterns; Insulin Sensitization; Glucose Intolerance; Intolerance
MeSH Terms: conditions — Heart Failure; Glucose Intolerance | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Avandia (Rosiglitazone)
Drug: Avanclia (Rosiqlitazone)

SUMMARY:
This study will evaluate the safety and effectiveness of the drug rosiglitazone for improving heart function in patients with heart failure and glucose intolerance or type II (adult-onset) diabetes, or both. Because of a lowered sensitivity to the hormone insulin, patients with type II diabetes or glucose-intolerance do not regulate glucose (sugar) effectively. Rosiglitazone is used to treat type II diabetes, but it is not commonly given to patients with heart failure because it can cause leg swelling and, rarely, pulmonary edema. However, patients with heart failure who also have glucose intolerance or type II diabetes generally fare worse than those with heart failure alone, and therapies that decrease insulin resistance may be beneficial to these patients.

Patients 21 years of age and older with heart failure and type II diabetes or glucose intolerance, or both, may be eligible for this study. Patients must be stable on current therapy for heart failure and must not have any planned surgeries for coronary artery disease. Candidates will be admitted to the NIH Clinical Center for from 2 to 7 days for screening procedures, which include a medical history and physical examination, blood and urine tests, electrocardiogram (ECG), chest x-ray, magnetic resonance imaging (MRI), exercise testing, and echocardiography (ultrasound test of the heart).

Participants will be randomly assigned to receive either rosiglitazone or placebo (an identical-looking pill with no active ingredient). They will take one tablet a day for the first month, one tablet twice a day for the second month, and then two tablets twice a day from the third month to the end of the study at 6 months. During the treatment period, patients will have a history, physical examination, and blood tests every 4 weeks, exercise testing and echocardiography at 3 and 6 months, and urinalysis, electrocardiogram and MRI at 6 months. To check for fluid accumulation in the legs or lungs, patients will report their weight and symptoms every 2 weeks throughout the study. After the 6-month treatment period, patients will be put back on the diabetes medicines they were taking before the study. Their physicians will be notified of possible modifications in treatment for maintaining optimum glucose tolerance.

Six months after completing treatment (one year after beginning the study), patients will return to the Clinical Center for blood tests to measure the long-term effects of rosiglitazone and to evaluate progress. They will then be invited to return to the clinic for annual checkups, if possible, or for yearly follow-up by mail or telephone to review their health status.

DETAILED DESCRIPTION:
The current medical management for heart failure invariably employs a 'one treatment fits all' approach. The failure to appreciate specific genotypic/phenotypic features in heart failure subjects is postulated to be a reason recent heart failure studies evaluating the efficacy of tumor necrosis factor alpha antagonists and endothelin receptor blockers showed no overall benefit. This experience suggests that the future improvement in the medical management of patients with heart failure may require pre-prescription genotyping/phenotyping to tailor drug therapy to the underlying mechanistic processes orchestrating the development and progression of heart failure.

In this regard, the insulin-resistance syndrome has been recognized as a significant associated factor with the development of cardiac hypertrophy and heart failure. A novel class of agents has been developed that increase insulin sensitivity via the activation of the transcription factor-peroxisomal proliferators activated receptor gamma (PPAR gamma). These drugs, known as the thiazolidinediones are currently licensed for the treatment of type II diabetes mellitus. Interestingly, at the preclinical level, PPAR gamma appears to play a regulatory role in attenuating the development of cardiac hypertrophy and thiazolidinedione therapy has been shown to attenuate the development of contractile dysfunction in mice following myocardial infarction.

The hypothesis intrinsic to this proposal is that insulin resistance is commonly associated with the development/progression of heart failure and that improving insulin sensitivity will be of clinical benefit in this select group of patients with heart failure. The primary objective of this study is to establish the safety and efficacy of thiazolidinedione therapy in insulin-resistant heart failure subjects. The study is designed as a phase II, randomized, double-blind, placebo-controlled dose escalation study. The primary outcomes will be the safety of administration, and the evaluation of the modulation in contractile function in heart failure subjects treated with thiazolidnediones. Moreover, changes in functional capacity and the determination of the biochemical and genomic modification of heart failure and insulin-resistance will be measured in response to thiazolidnedione therapy in heart failure subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult normal volunteers, age matched (55-75 years of age)

Adult patients greater than 21 years of age who meet the following criteria:

* Heart Failure due to ischemic heart disease or of idiopathic etiology
* Depressed LV systolic function, EF less than or equal to 0.45 by Radionuclide Angiography (MUGA)
* New York Heart Association Functional Class II or III
* Patient stable on current heart failure therapy
* Evidence of insulin resistance or type II diabetes on insulin-sensitivity screening
* No predicted cardiac revascularization therapy requirements

EXCLUSION CRITERIA:

Pregnant or lactating

History of admission for acute heart failure exacerbation within last one month

Acute myocardial infarction within the last three months

Cardiac resynchronization pacemaker placement within the last three months

Genetic defect known to have induced heart failure

Serum creatinine greater than 2.5 mg/dL.

Liver transaminase levels greater than 2.5 x upper limit of normal

Requirement for insulin therapy to control blood glucose

Current use of thiazolidinedione for diabetic control or history of discontinuation of thiazolidinedione therapy following development of side effects

Uncontrolled blood glucose levels or the use of insulin therapy to control diabetes

Immune compromise including chronic HIV, HBV, and HCV infection

Chronic systemic inflammatory disease such as SLE, rheumatoid arthritis, collagen vascular disease

Participation in unrelated research involving investigational pharmacological agent 30 days before planned dosing

Current alcohol or drug abuse

Inability to provide informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-07-09; Study Completion 2007-04-11

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Heart, Lung and Blood Institute (NHLBI), 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Coats AJ. Angiotensin type-1 receptor blockers in heart failure. Prog Cardiovasc Dis. 2002 Jan-Feb;44(4):231-42. doi: 10.1053/pcad.2002.31585. PMID 12007079